CLINICAL TRIAL: NCT03853031
Title: Transesophageal Echocardiology Measured Left Ventricular End Diastolic Area (LVEDA) As Guide for Fluid Therapy in Major Oncosurgeries
Brief Title: Transesophageal Echocardiology Measured Left Ventricular End Diastolic Area As Guide for Fluid Therapy in Major Oncosurgeries
Acronym: TEE LVEDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr Anita Kulkarni, Principal Investigator, Rajiv Gandhi Cancer Institute & Research Center, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RGCIRC Rohini
Record Dates: First submitted 2019-02-08; First posted 2019-02-25 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Fluid Therapy DURING SURGERY
Keywords: Fluid therapy; Left ventricular end diastolic area; Central venous pressure
MeSH Terms: interventions — COP protocol 2; Control Groups

STUDY DESIGN:
Intervention Model Description: During surgery Control group of patients will receive CVP guided fluids Study group of patients will receive TEE measured LVEDA guided fluids
Who Masked: Participant
Masking Description: Patients will be randomly allotted to either TEE or CVP Group according to computer generated randomization thus will be masked .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LVEDA guided intraoperative fluid therapy (Active Comparator): Patients in TEE group will be given crystalloid fluids during surgery guided by LVEDA cm2 to be maintained between 10 -18 cm2 , if LVEDA < 10 cm2 then 200ml colloid bolus will be given and increase in LVEDA noted.
  Interventions: Procedure: LVEDA cm2 guided intraoperative fluid in TEE /Study Group
- CVP guided intraoperative fluid therapy (Active Comparator): Patients in CVP group will be given crystalloid fluids during surgery guided by CVP values to be maintained between 10 -16 cms of water H2O ,if CVP value < 10 cms H2O then 200 ml colloid bolus will be given and increase in CVP value noted.
  Interventions: Procedure: CVP guided intraoperative fluid in CVP / Control group

INTERVENTIONS:
Procedure: LVEDA cm2 guided intraoperative fluid in TEE /Study Group — Placement of Transoesophageal echocardiography probe in TEE group to measure Left ventricular end diastolic area cm2
  Arms: LVEDA guided intraoperative fluid therapy
Procedure: CVP guided intraoperative fluid in CVP / Control group — Ultrasound guided Internal Jugular Vein catheter placement in CVP group to measure CVP value cms H2O .
  Arms: CVP guided intraoperative fluid therapy

SUMMARY:
Intraoperative fluid management is pivotal to successful outcome of major oncosurgeries . Adequate volume replacement to achieve optimal cardiac performance is critical to prevent any deleterious consequences of under resuscitation or fluid overload . Traditionally CVP monitoring has been tool to guide intraoperative fluid therapy and has poor reliability as indicator of volume status . Transesophageal Echocardiography measured LVEDA is more reliable and sensitive measure of left ventricular volume to guide intraoperative fluid therapy . Investigators plan the study comparing total fluid requirement and postoperative outcomes in two groups of patients receiving central venous pressure (CVP) guided Conventional Fluid Therapy (CFT) and Left ventricular end diastolic area( LVEDA) guided fluids for major oncosurgeries.

DETAILED DESCRIPTION:
Adult patients undergoing major oncosurgeries will be included in the study ,with Alpha Error(%) = 5 ,Power(%)= 80 ,required sample size per group is 29.Investigators will include 30 patients in each group. Patients will be randomly allotted to Central Venous Pressure CVP Group (Control Group) or Transesophageal Echocardiography TEE Group (Study Group) according to computer generated randomization. In the OR 5 lead Electrocardiogram ( ECG ), Oxygen saturation (SPO2 ), Noninvasive blood Pressure (NIBP) , End tidal carbon di oxide (ETCO2 )monitors will be attached .Under local anesthesia 16Gauge peripheral intravenous and Radial artery cannulation will be performed . Anesthesia will be induced with Fentanyl 1mcg/kg-1, Morphine 0.05mg/kg-1, Propofol titrated dosage 1-2 mg/kg-1 and neuromuscular blockade with Atracurium 0.5mg/kg-1.Trachea will be intubated with oral cuffed endotracheal tube of appropriate size. Anaesthesia will be maintained with O2 / Air mixture 40:60 % Intermittent Positive Pressure Ventilation with Sevoflurane , intermittent boluses of Fentanyl and Train of Four ratio guided Atracurium . Postintubation ultrasound guided internal jugular vein will be cannulated with B.Braun 7French 20cm, 16 G Triple lumen central venous catheter in both CVP and TEE Group patients . My Lab Five ESAOTE TEE 022 multiplane probe ,frequency 3 to7MHz (Providian Medical Equipment ,OH) will be placed in TEE Group patients.Intraoperative all patients will be given one-third starvation fluid in first hour of surgery , maintenance fluid 2ml/hour crystalloid . Target is to maintain CVP between 10 -16 cms of water (H20) in CVP Group , values will be recorded every 30 minutes if CVP decreases < 10 then 200 ml colloid bolus will be given and increase in CVP value noted . In the TEE Group TEE probe will be inserted in the oesophagus (40-45 cms) adjusted to obtain mid-papillary transgastric short axis view ,the desired view will be freezed at end-diastole and the left ventricular cavity will be traced including the papillary muscles to obtain left ventricular end diastolic area in cm2 , the average of three readings at particular interval will be noted . Every half hourly values will be measured and also if systolic blood pressure < 90 mm Hg . Fluid therapy will be given with the target to maintain LVEDA ≥ 10 cm2 (ranging between 10-18 cm2). For readings < 10 cm2 colloid bolus 200 ml will be given and increase in the LVEDA will be noted.For same readings Left Ventricular Outflow trac ( LVOT) view will be obtained to measure aortic diameter at the cusps and LVOT VTI , Stroke volume ( SV) will be calculated as LVOT area { Pi (LVOT diameter /2 } 2 × LVOT VTI and Cardiac Outpt will be calculated as SV x Heart Rate . Increase in stoke volume and cardiac output with colloid boluses will be noted.Urine output will be recorded every 30 minutes in all the patients.Titrated noradrenaline infusion (conc 0.08mg/ml ) will be started if Mean Arterial Pressure (MAP) < 70 mmHg with optimal fluid administration in CVP and TEE group .Serum lactate levels will be measured on completion of surgery and postoperative at 24 and 48 hours, neuromuscular blockade will be reversed and trachea extubated . In PACU both groups will receive CVP guided intravenous fluids, monitoring will include heart rate , Blood Pressure ,SPO2 , CVP , urine output. Note will be made of any patient requiring postoperative ventilator support, inotropic support,return of bowel sounds, serum lactate levels and serum creatinine levels at 24 and 48 hours and length of ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing major abdominopelvic oncosurgeries .

Exclusion Criteria:

* oesophageal varices
* carcinoma oesophagus
* carcinoma stomach
* coagulopathies
* duration of surgery exceeding 8 hours.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
To calculate total intraoperative fluids required in TEE (study) and CVP (control) groups. | Upto 8 hours
  During the surgery Study group will receive fluids ( crystalloids and bolus colloids) guided by LVEDA cm2 and Control group will receive fluids (crystalloids and bolus colloids) guided by CVP cms H20

SECONDARY OUTCOMES:
To compare serum lactate levels in millimols/litre | upto 48 hours
  In both the groups through completion of surgery and at postoperative 24 hours and postoperative 48 hours serum lactate levels will be measured .
To compare serum creatinine in milligrams per decilitre in both the groups | Upto 48 hours.
  In both groups serum creatinine in milligrams per decilitre will be measured at postoperative 24 and postoperative 48 hours.
Length of ICU stay | Upto 10 days
  In both the groups postoperative stay in the ICU will be noted in days.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kulkarni, MD, Principal Investigator — Rajiv Gandhi Cancer Institute & Research Centre , India; Anita Kulkarni, M.D., Principal Investigator — Rajiv Gandhi Cancer Institute & Research Centre , India
Locations (1):
- Anita Kulkarni, Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gutierrez MC, Moore PG, Liu H. Goal-directed therapy in intraoperative fluid and hemodynamic management. J Biomed Res. 2013 Sep;27(5):357-65. doi: 10.7555/JBR.27.20120128. Epub 2013 Mar 10. PMID 24086168
- [Background] Cheung AT, Savino JS, Weiss SJ, Aukburg SJ, Berlin JA. Echocardiographic and hemodynamic indexes of left ventricular preload in patients with normal and abnormal ventricular function. Anesthesiology. 1994 Aug;81(2):376-87. doi: 10.1097/00000542-199408000-00016. PMID 8053588
- [Background] Marik PE, Cavallazzi R. Does the central venous pressure predict fluid responsiveness? An updated meta-analysis and a plea for some common sense. Crit Care Med. 2013 Jul;41(7):1774-81. doi: 10.1097/CCM.0b013e31828a25fd. PMID 23774337